CLINICAL TRIAL: NCT04975763
Title: Dietary Oils to Sustain Energy (DOSE) Study: Understanding How Consumption of Dietary Oils in Foods Influences Blood Fatty Acids and Body Weight
Brief Title: Dietary Oils to Sustain Energy Study
Acronym: DOSE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Martha Belury, Associate Professor, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021H0232
Record Dates: First submitted 2021-07-15; First posted 2021-07-23 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Soybean Oil (Experimental): Consumption of study foods each day made with soybean oil
  Interventions: Other: Soybean Oil Foods
- Palm Oil (Placebo Comparator): Consumption of study foods each day made with palm oil
  Interventions: Other: Palm Oil Foods

INTERVENTIONS:
Other: Soybean Oil Foods — Three food product containing 10g of soybean oil each will be consumed each day for a today of 30g of soybean oil consumed each day
  Arms: Soybean Oil
Other: Palm Oil Foods — Three food product containing 10g of palm oil each will be consumed each day for a today of 30g of palm oil consumed each day
  Arms: Palm Oil

SUMMARY:
The research study is an intervention and feasibility crossover design pilot study designed to assess if consuming 3 study foods made with either soybean oil or palm oil per day for 4 weeks can alter whole blood, plasma and erythrocyte fatty acids and body weight in overweight/obese adults. Additionally, the study will assess the adherence to consuming 3 study foods per day for 4 weeks and to assess if participant remain unaware of (or masked to) which study food group (soybean oil vs palm oil) they are consuming.

DETAILED DESCRIPTION:
The objectives of the study include

* To determine changes in whole blood, plasma and erythrocyte linoleic acid after 4 weeks of consuming 3 foods products made soybean oil and determine changes in plasma and erythrocyte oleic acid and palmitic acid after 4 weeks of consuming 3 food products per day made with palm oil in overweight/obese adults
* To determine changes in body weight in overweight/obese adults during four weeks of consuming 3 food products per day made with soybean oil and during four weeks of consuming 3 food products per day made with palm oil
* To determine if there is evidence of unmasking of the two food product groups (soybean oil or palm oil) during the study in participants and in study coordinators
* To determine adherence of consuming 3 food products per day made with either soybean or palm oil for 4 weeks in overweight/obese adults

ELIGIBILITY:
Inclusion Criteria:

* Age 25-80 years old
* Nonsmokers
* BMI 25-55 kg/m2

Exclusion Criteria:

* Current or previous diagnosis of heart, kidney, and some liver diseases
* Current or previous diagnosis some circulatory diseases and some autoimmune diseases
* Treatment of current cancer diagnosis or current cancer diagnosis
* Current or previous diagnosis of diabetes
* Gastrointestinal diseases or disorders (including pancreatic) that influence nutrient digestion and absorption or gastric bypass surgery
* Alcohol or drug abuse
* Inability to access veins for venipuncture
* Hypothyroidism or Hyperthyroidism diagnosis
* Food Allergy or intolerances
* Any dietary restriction where consumption of the study foods or any ingredient would be contraindicated
* Use of medications where consuming the study foods would be contraindicated
* Use of supplements or medications for weight loss or following a weight loss program
* Use of supplements high in linoleic acid in the past 4 weeks prior to enrolling
* Pregnancy and lactation

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-07-19 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in blood fatty acid composition | Week 0, Week 2, Week 4, Week 6, Week 8, Week 10
  Determine changes in whole blood, plasma and erythrocyte linoleic acid in the soybean oil arm and determine the changes in whole blood, plasma and erythrocyte oleic acid and palmitic acid in the palm oil arm. Fatty acids for all sample types are reported as percent of total identified

SECONDARY OUTCOMES:
Changes in body weight | Week 0, Week 2, Week 4, Week 6, Week 8, Week 10
  Determine changes in body weight in the soybean oil and palm oil arms
Evidence of unmasking | Week 4 and Week 10
  Determine if there is evidence of unmasking of the two food product groups (soybean oil or palm oil) during the study in participants and in study coordinators using a questionnaire and calculating the Bang Blinding Index scale ranging from -1 to 1 with -1 is opposite guessing, 1 is lack of blinding and 0 is blinding
Adherence to study food consumption | Week 2, Week 4, Week 8, Week 10
  Determine adherence of consuming 3 food products per day made with either soybean or palm oil through self report and returning of uneaten foods

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Human Nutrition Laboratory, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cole RM, Colombo E, Angelotti A, Sparagna GC, Choriego RE, Jimenez-Flores R, Ni A, Belury MA. Feasibility Study of Soybean Oil-Fortified Foods to Alter Blood Content of Linoleic Acid and Body Weight: A Randomized Double-Masked Placebo-Controlled Crossover Trial. J Nutr. 2025 Dec 27:101288. doi: 10.1016/j.tjnut.2025.101288. Online ahead of print. PMID 41461275